CLINICAL TRIAL: NCT03440229
Title: Functional Research of Emulsifiers in Humans
Acronym: FRESH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Georgia State University (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, James Lewis, Professor of Medicine, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 828422; R21DK115180 (NIH)
Record Dates: First submitted 2018-02-05; First posted 2018-02-22 (Actual); Results first posted 2021-09-16 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-09

CONDITIONS: Healthy
MeSH Terms: interventions — Carboxymethylcellulose Sodium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a randomized double-blind controlled feeding experiment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Emuslfier-free diet (No Intervention): This is western style diet prepared without any emulsifiers. Emulsifier free brownies and sorbet are provided daily.
- Emulsifier-containing diet (Experimental): This is a western style diet prepared without any emulsifiers with the exception of the CMC that is included in brownies and sorbet that are provided daily.
  Interventions: Other: Emulsifier-containing diet

INTERVENTIONS:
Other: Emulsifier-containing diet — CMC is one of many synthetic dietary emulsifiers that are incorporated into a variety of processed foods. We have recently shown that, in mice, consumption of P80 and CMC, alters microbiota composition, have pro-inflammatory potential and promote microbiota encroachment into the colonic mucosa, low-grade inflammation, and metabolic syndrome. However, it is not known whether these compounds have similar effects in humans. We would like to study these effects in the human gut microbiota.
  Other Names: Carboxymethylcellulose (CMC)
  Arms: Emulsifier-containing diet

SUMMARY:
A randomized double-blind study of the effect of carboxymethylcellulose (CMC) on stool microbiota composition, microbiota localization, and metabolic parameters in healthy subjects. It includes a 11-day in-patient stay, randomization to an emulsifier-free group or a CMC group with the same diet except baked goods/sorbet with added CMC at 15g/person/day.

DETAILED DESCRIPTION:
This is a randomized double-blind, controlled feeding experiment examining the effect of CMC on the stool microbiota composition, gene expression, and microbiota localization with respect to the epithelium. In addition, the investigators will assess the impact of CMC exposure in the diet on markers of metabolic syndrome including response to oral glucose tolerance testing and other plasma metabolite measurements.

Sixteen healthy volunteers were be recruited. 3 were admitted for 17 days and 13 participants were admitted for an 11-day in-patient study. All participants received 3 full days of freshly prepared emulsifier-free food to begin the study. This will be called the "washout period". Those will a 17 day stay received the wash out diet while inpatient and those with an 11 day stay received the wash out dies while out patient. Participants will then be randomized into an "emulsifier-free" arm and a "CMC" arm in a 1:1 ratio. Both arms will continue the same diet except that the "CMC" arm's brownie and sorbet will have CMC added to achieve a level of 15 gm per person per day consumption. Serial collection of fecal, plasma, urine and mucosal biopsy samples will be performed to investigate the extent to which CMC consumption by humans impacts the gut microbiota and its interaction with the host parameters related to inflammation and metabolism. Participants will have daily urine and stool collections. Sigmoidoscopies and glucose tolerance testing will be completed on the day prior to the start of the intervention and the last day of the inpatient stay (Days 4 and 17 for the 3 participants with a 17 day stay and days 1 and 11 for participants with an 11 day stay. Blood samples were collected on days 1-4, 5, 8, 10, 12, 15, and 17 for those with a 17 day inpatient stay and 1-4, 8, 10, and 11 for those with an 11 day stay.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is capable of giving informed consent
2. Participant is age 18 to 60 years

Exclusion Criteria:

1. Diagnosis with Inflammatory Bowel Disease (IBD), celiac disease, or other chronic intestinal disorders. Since we are interested in assessing the impact of diet on the microbiome in the absence of pathologic inflammation, we will exclude participants with chronic intestinal abnormalities.
2. Baseline bowel frequency less than every 2 days or greater than 3 times daily. Normal bowel frequency is every 3rd day to 3 times per day.20-23 Although unknown, stool frequency could be related to the microbiome composition.24-26 Furthermore, change in diet could alter baseline stool frequency, potentially causing diarrhea, particularly in those with high baseline stool frequency, or severe constipation in those with low stool frequency. To avoid the need for use of antidiarrheal medications or laxatives, which themselves could alter the microbiome composition, these patients will be excluded.
3. Current smoker. What effect smoking has on the microbiome of the gut is unknown. Furthermore, because our hospital is a smoke-free environment, volunteers will not be able to smoke. Thus, inclusion of smokers would increase the risk of early withdrawal from the study.
4. Body Mass Index (BMI) <18.5 or >40 at screening. Volunteers with BMI below normal27 will be excluded to prevent inclusion of participants with a subclinical systemic disease that may influence the gut microbiome. Volunteers with severe obesity will be excluded as obesity may be associated with altered gut microbiome composition.
5. More than two of the criteria for metabolic syndrome:

   * A waist circumference greater than 35 inches (89 centimeters) for women and 40 inches (102 centimeters) for men at screening.
   * A diagnosis of diabetes mellitus or baseline HbA1c > 6.4% or a fasting glucose level of greater than 100mg/dL
   * Systolic blood pressure >130 mmHg or diastolic blood pressure >85 mmHg or treated with medications for hypertension at screening.
   * Fasting triglycerides >149 mg/dl or treated with medications for hypertriglyceridemia
   * Fasting HDL cholesterol <40 mg/dl in men or <50 mg/dl in women or treated with medications for hypercholesterolemia
6. Known substance abuse disorder or consumption of illicit drugs or alcohol in the 24 hours prior to admission to the Center for Human Phenomic Science (CHPS).
7. Prior bowel resection surgery other than appendectomy. It is unknown how prior bowel resection surgery may influence the microbiome composition, hence we will exclude these participants.
8. Contraindication to flexible sigmoidoscopy and biopsies. Patients with suppressed white blood count may be at increased risk of systemic infection following sigmoidoscopy with biopsies. As such, participants with a white blood cell (WBC) less than 3,500 or an absolute neutrophil count of less than 1,000 will be excluded. Patients with thrombocytopenia or with a coagulopathy may be at increased risk of bleeding complications after colonoscopic biopsies. As such, patients with a platelet count of less than 100,000 or an international normalized ratio (INR) greater than 1.2 will be excluded from the study.
9. Estimated glomerular filtration rate (GFR)<60ml/min/1.73m2 based on measured serum creatinine concentration
10. Pregnant and lactating women. To avoid any risk to an unborn fetus or new born baby from changing the mother's diet, pregnant and lactating women will be excluded.
11. Use of antibiotics in the 6 months prior to Visit 2. A small proportion of bacteria may require 6 months to recover after treatment with antibiotics.28
12. Use of antacids, NSAIDs, or dietary supplements in the week prior to Visit 2. NSAIDs have been associated with C. difficile colitis, although whether this is causative and whether this is mediated through changing the fecal microbiota composition is unknown.29 Antacids could potentially alter the gut microbiota by changing the acid milieu or by altering fecal transit time. For our study purposes, multivitamins will not be considered dietary supplements.
13. Use of laxatives or anti-diarrhea medications in the two weeks prior to Visit 2.
14. Use of anticholinergics in the week prior Visit 2.
15. Use of narcotics in the week prior to Visit 2.
16. HIV infection, AIDS, or other known conditions resulting in immunosuppression - we will determine this by direct participant query; no formal testing will be done.
17. Allergies or intolerance to the components of the study diets.
18. Participant has experienced diarrhea within the two weeks prior to Visit 2. Diarrhea is defined as a change in bowel habits with an increased frequency or loose stools such that the stool could not be lifted with a fork.
19. Refusal to use a medically accepted method of birth control while participating in this study, such as a barrier method, hormonal contraceptives, implanted birth control devices, permanent methods (such as a vasectomy), and/or abstinence.
20. Vegans and Vegetarians.
21. Student or employee of any one of the investigators.
22. Anyone who cannot receive study payment (ie: visa)
23. Any condition that the investigator feels may limit the volunteer's ability to complete the study protocol.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2018-04-06 (Actual); Primary Completion 2019-05-13 (Actual); Study Completion 2019-05-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jim Lewis, MD, MSCE, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Doucet E, Pomerleau M, Harper ME. Fasting and postprandial total ghrelin remain unchanged after short-term energy restriction. J Clin Endocrinol Metab. 2004 Apr;89(4):1727-32. doi: 10.1210/jc.2003-031459. PMID 15070937
- [Derived] Chassaing B, Compher C, Bonhomme B, Liu Q, Tian Y, Walters W, Nessel L, Delaroque C, Hao F, Gershuni V, Chau L, Ni J, Bewtra M, Albenberg L, Bretin A, McKeever L, Ley RE, Patterson AD, Wu GD, Gewirtz AT, Lewis JD. Randomized Controlled-Feeding Study of Dietary Emulsifier Carboxymethylcellulose Reveals Detrimental Impacts on the Gut Microbiota and Metabolome. Gastroenterology. 2022 Mar;162(3):743-756. doi: 10.1053/j.gastro.2021.11.006. Epub 2021 Nov 11. PMID 34774538

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were 29 participants who were consented to the study. 8 were found to be ineligible prior to being randomized, 5 additional participants withdrew prior to being randomized saying they were no longer interested or able to participate and 16 participants were randomized.
Period: Overall Study
Arm/Group | Emuslfier-free Diet | Emulsifier-containing Diet
Started | 9 | 7
Completed | 9 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Emuslfier-free Diet | Emulsifier-containing Diet | Total
Number analyzed (Participants) | 9 | 7 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.11 (12.72) | 35.24 (11.28) | 38.54 (12.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 9
  Male | 3 | 4 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 3 | 9
  White | 3 | 2 | 5
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Height [Mean (Standard Deviation); unit: cm] | 170.01 (12.36) | 168.22 (6.91) | 169.23 (10.07)
Weight [Mean (Standard Deviation); unit: kg] | 69.58 (13.16) | 70.64 (10.63) | 70.05 (11.74)
BMI [Mean (Standard Deviation); unit: kg/m2] | 24.06 (3.62) | 25.02 (3.88) | 24.48 (3.64)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 115.33 (8.53) | 124.71 (9.12) | 119.44 (9.76)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 69.78 (14.06) | 71.86 (8.17) | 70.69 (11.55)

OUTCOME MEASURES:

1. Primary Outcome: Distance of Nearest Bacteria to the Epithelium
Description: Measured distance from the epithelium to the nearest bacteria under high powered microscopy; The measurements were taken on the last day of the diet intervention. An average of 3 measurements was taken.
Time Frame: last day of inpatient stay (either day 17 for the 3 participants with a 17 day inpatient stay or day 11 for the 13 participants with an 11 day inpatient stay.)
Measure: Mean (Standard Deviation); unit: µm
Arm/Group | Emuslfier-free Diet | Emulsifier-containing Diet
Number analyzed (Participants) | 9 | 7
µm | 17.06776 (5.949757) | 14.09342 (12.51437)

2. Secondary Outcome: Change in Weight
Description: Comparison of weight change during the study period - pre and post intervention. Weight on the last day of the inpatient stay was substracted from weight after the washout period but before the start of the intervention.For 3 participants with a 17 day stay, weight from day 4 of the inpatient stay was substracted from day 17. For 13 with an 11 day stay, weight from Day 1 of the inpatient stay was substracted from Day 11
Time Frame: For 3 participants with a 17 day stay, weight was measured on Day 4 and Day 17 of the inpatient stay. For 13 participants with an 11 day stay, weight was measured on Day 1 and Day 11 of the inpatient stay.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Emuslfier-free Diet | Emulsifier-containing Diet
Number analyzed (Participants) | 9 | 7
kg | -1.341 (1.408) | -0.8111 (1.228)

3. Secondary Outcome: Area Under Glucose Concentration Curve
Description: Area under the glucose concentration curves during the oral glucose tolerance test. These measurements were obtained by subtracting the pre from the post net incremental area under the curve. For 3 participants with a 17 day stay, area under the glucose curve from day 4 of the inpatient stay was substracted from day 17. For 13 participants with an 11 day stay, area under the glucose curve from Day 1 of the inpatient stay was substracted from Day 11
Time Frame: For 3 participants with a 17 day stay, area under the glucose curve was measured on days 4 and 17 of the inpatient stay . For 13 participanst with an 11 day stay, area under the glucose curve was measured on days 1 and Day 11 of the inpatient stay.
Measure: Mean (Standard Deviation); unit: μIU*min/mL
Arm/Group | Emuslfier-free Diet | Emulsifier-containing Diet
Number analyzed (Participants) | 9 | 7
μIU*min/mL | -726.5 (1482.9) | -669.6 (1454.8)

4. Secondary Outcome: Area Under Insulin Concentration Curve
Description: Area under the insulin concentration curves during the oral glucose tolerance test. These measurements were obtained by subtracting the pre from the post net incremental area under the curve. This is measured in microliter international units/milliliter. For 3 participants with a 17 day stay, area under the insulin concentration curve from day 4 of the inpatient stay was substracted from day 17. For 13 participants with an 11 day stay, area under the insulin concentration curve from Day 1 of the inpatient stay was substracted from Day 11
Time Frame: For 3 pts. with 17 day stays, area under the curve was measured on days 4 and 17 of the inpatient stay. For 13 pts. with 11 day stays, area under the curve was measured on days 1 and Day 11 of the inpatient stay.
Measure: Mean (Standard Deviation); unit: μIU*min/mL
Arm/Group | Emuslfier-free Diet | Emulsifier-containing Diet
Number analyzed (Participants) | 9 | 7
μIU*min/mL | -1325.4 (1444.6) | 1506.4 (2756.2)

5. Secondary Outcome: Visual Analog Scale Measurements - Satiety/Hunger - Change From Baseline
Description: Desire to eat, hunger, fullness, and prospective food consumption were rated on a 150-mm visual analog scale (VAS) that was adapted from Hill and Blundell in Doucet et al.(see references) The Satiety questionnaire was given before a meal (preprandial) and after the meal (postprandial). The minimum score is 0mm and the maximum score is 150mm for each question. The score prior to the intervention was subtracted from the post intervention score measured on the last day of the inpatient stay. Each question is scored individually. Higher score means more of the characteristic being measured. There are no better or worse outcomes based on these scores.
Time Frame: Measured at end of inpatient stay (Day 17 for 3 participants and Day 11 for 13 participants) comparing it to the study start (prior to diet intervention; either day 4 for the 3 participants or day 1 for 13 participants.
Population: One participant on the emulsifier free diet did not answer the last 3 question on the Satiety and Hunger questionnaire.
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Emuslfier-free Diet | Emulsifier-containing Diet
Number analyzed (Participants) | 9 | 7
millimeters
  How hungry do you feel? (pre-prandial at study end minuse pre-prandial at study start) | 10.778 (62.036) | -6.714 (23.365)
  How full do you feel? (Post-prandial at study end minus post-prandial at study start) | -17.444 (41.564) | -12.571 (31.989)
  How strong is your desire to eat? (Pre-prandial at Study End Minus pre-prandial at Study Start) | -9.889 (45.460) | 2.857 (31.583)
  How much do you think you could eat now? (Preprandial at Study End Minus preprandial at Study Start): number analyzed (Participants) | 8 | 7
  How much do you think you could eat now? (Preprandial at Study End Minus preprandial at Study Start) | -18.375 (46.986) | -0.286 (47.328)
  Urge to eat? (Pre-prandial at Study End Minus Pre-prandial at Study Start): number analyzed (Participants) | 8 | 7
  Urge to eat? (Pre-prandial at Study End Minus Pre-prandial at Study Start) | 7.750 (18.235) | -9.571 (42.442)
  Urge to eat? (Post-prandial at Study End Minus Post-prandial at Study Start): number analyzed (Participants) | 8 | 7
  Urge to eat? (Post-prandial at Study End Minus Post-prandial at Study Start) | 18.778 (41.355) | 7.429 (22.948)
  Preoccupation with thoughts of food (Pre-prandial at Study End Minus Pre-prandial at Study Start): number analyzed (Participants) | 8 | 7
  Preoccupation with thoughts of food (Pre-prandial at Study End Minus Pre-prandial at Study Start) | 12.375 (33.781) | -7.000 (43.420)
  Preoccupation with thoughts of food (Post-prandial at Study End Minus Post-prandial at Study Start): number analyzed (Participants) | 8 | 7
  Preoccupation with thoughts of food (Post-prandial at Study End Minus Post-prandial at Study Start) | 31.667 (39.138) | 15.857 (24.341)

6. Secondary Outcome: Fecal Lipocalin-2
Description: Fecal lipocalin-2 by Elisa
Time Frame: For the 3 participants with a 17 day inpatiet stay, this was measured on Day 17. For the 13 participants with an 11 day stay, this was measured on Day 11
Measure: Mean (Standard Deviation); unit: ng/gm
Arm/Group | Emuslfier-free Diet | Emulsifier-containing Diet
Number analyzed (Participants) | 9 | 7
ng/gm | 588.9959 (180.832) | 304.3584 (101.7004)

ADVERSE EVENTS:
Time Frame: Participants were asked about adverse events at each visit starting at the screening visit and through the last visit. This is approximately 164 days.
Description: At screening, participants were asked about any symptoms they were currently experiencing. Participants were asked at each subsequent visit whether they experienced any AEs since the last visit. They were also asked if previously reported unresolved AEs had resolved. The start/end dates were recorded for each AE along with severity (grade), relatedness to study intervention, and whether any action was taken with the study intervention (i.e. paused intervention, stopped intervention)
Arm/Group | Emuslfier-free Diet | Emulsifier-containing Diet
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/7
Other Adverse Events (participants affected / at risk) | 3/9 | 1/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Emuslfier-free Diet (N=9) | Emulsifier-containing Diet (N=7)
Headache (General disorders) | 2 (2) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-14): https://cdn.clinicaltrials.gov/large-docs/29/NCT03440229/Prot_SAP_000.pdf